CLINICAL TRIAL: NCT00202891
Title: Sisomicin Cream Vs Nadifloxacin Cream in Primary Pyodermas
Brief Title: Sisomicin Cream Vs Nadifloxacin Cream in Primary Pyodermas (Study P04460)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No further local interest in pursuing the study.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Fulford India Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04460
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Pyoderma
Keywords: pyoderma; sisomicin; nadifloxacin
MeSH Terms: conditions — Pyoderma | interventions — Sisomicin

INTERVENTIONS:
Drug: sisomicin

SUMMARY:
This open-label, randomized, parallel-group clinical study is designed to compare the efficacy and safety of the topical antibiotic, sisomicin cream, with that of another topical antibiotic cream, nadifloxacin cream, in the treatment of Indian patients with primary pyodermas.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and suffering from primary pyodermas requiring topical antibiotic therapy without occlusive dressings.
* >=6 years of age.
* Written informed consent.

Exclusion Criteria:

* Patients must not take any other antibiotics.
* Patients should not be hypersensitive to any of the test drugs.
* Patients are not to have any other investigational drug within one month of starting this study.
* Patients cannot be enrolled more than once in the study.
* Patients must not have any significant medical condition which, in the judgment of the investigator, might interfere with the study or require treatment.
* Pregnant women and nursing mothers are to be excluded.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Study Completion 2007-09 (Actual)